CLINICAL TRIAL: NCT05983055
Title: Suitability of Periarticular Steroid Injections for Sickle Cell Arthropathy Pain Therapy
Brief Title: Steroid Injection for Sickle Cell Arthropathy Pain Therapy
Status: Completed | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAn2018 SCD arthro injectn
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; Sickle Cell Abnormality
Keywords: Sickle cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dexamethasone 20mg — Periarticular dexamethasone injection
  Other Names: Dexamethasone injection

SUMMARY:
Sickle cell disease (SCD) is associated with arthropathy. Arthropathy may require periarticular corticosteroid injection therapy. This observational study examines efficacy, and safety of steroid injections in SCD patients. Data collection includes patient's gender, age, race, smoking history, alcohol intake, analgesic use, pain score, sleep quality, limb joint injections, post-injection analgesia, and post-injection complication. Pain is measured using numeric pain scale. Sleep quality is measured using Likert scale.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is associated with arthropathy. Arthropathy causes pain which may require periarticular corticosteroid injection therapy. There is inadequate data about the suitability of steroid therapy in SCD patients. This prospective observational study examines the efficacy, and safety of periarticular steroid injections in SCD patients.

This is a cohort study of adult patients undergoing pain management at a pain clinic in Canada. Data collection includes patient's gender, age, race, smoking history, alcohol intake, analgesic usage, numeric pain score, sleep quality score, limb joint injections, post-injection analgesia, and post-injection complication. Pain is measured using numeric pain rating scale. Sleep quality is measured using the Likert Sleep scale. A change in the pain or sleep scores by 2-points is considered significant. Data are analyzed with IBM® SPSS® Statistics 25; using Student's t-test, ANOVA, Pearson Chi-square test, and regression analysis. P-value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients
* sickle cell disease arthropathy
* periarticular steroid injection therapy
* regular sleep diary
* regular pain diary
* informed consent for therapy and diary review

Exclusion Criteria:

* pediatric patients
* patient without sickle cell disease arthropathy
* patient without periarticular steroid injection
* irregular sleep diary
* irregular pain diary

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of consecutive adult patients who underwent pain management at a pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Numeric pain score, objective measurement using validated Numeric Pain Rating scale | 12 weeks
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

SECONDARY OUTCOMES:
Sleep quality score, objective measurement using validated Likert sleep scale | 12 weeks
  Sleep quality score, using the Likert sleep scale of 0 to 10, low scores indicate poor sleep, high scores indicate better sleep

CONTACTS AND LOCATIONS:
Overall Officials: Olumuyiwa Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No